CLINICAL TRIAL: NCT05864352
Title: The Role of Dietary Titanium Dioxide on the Human Gut Microbiome and Health
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Lowell (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency); Wright Labs (Unknown)
Responsible Party: Principal Investigator, Kelsey Mangano, Associate Professor, University of Massachusetts, Lowell
Other Study IDs: 21-122-MAN-XPD
Record Dates: First submitted 2023-05-08; First posted 2023-05-18 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Inflammation; Microbiota; Gastrointestinal Irritation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Three consecutive fecal samples frozen at -80 degrees C
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High TiO2 Consumer: Participants with an estimated TiO2 stool content greater than the cohort median content, μg/mg dry stool.
- Low TiO2 Consumer: Participants with an estimated TiO2 stool content less than the cohort median content, μg/mg dry stool.

SUMMARY:
This proposal will quantify dietary exposure of a nano- food additive in the U.S. food supply, and determine its impact on the human gut microbiome, gut inflammation, permeability and oxidative stress. Titanium dioxide (TiO2, or E171 food grade additive) is used in processed foods, with thousands of tons produced annually and an expected increase >8.9% from 2016 to 2025. Preclinical models demonstrate >99% of consumed TiO2 is retained within the intestinal lumen and excreted in the feces. In animal models, dietary TiO2 causes shifts in the gut microbiome, decreases acetate production, increases biofilm formation, and causes profound disruption of gut homeostasis and intestinal tight junctions, due to the production of reactive oxygen species and increased inflammation. However, the relation between chronic TiO2 intake and human gut homeostasis has yet to be elucidated. France issued an executive order to ban food grade TiO2 use after January 1st 2020, over serious safety concerns. Since then, multiple European civil societies have jointly called for an executive order to ban TiO2 across the EU. Typical TiO2 intake among U.S. adults remains to be documented, and there are no known studies that estimate dietary exposure of TiO2 using a whole foods approach. Therefore, the overarching goals of this project are to: 1) measure dietary TiO2 exposure in a sample of U.S. adults, using dietary recalls and fecal TiO2 content; 2) determine how fecal TiO2 content is related to gut dysbiosis, metatranscriptomics, intestinal inflammation, permeability and oxidative stress.

DETAILED DESCRIPTION:
The U.S. food supply contains large amounts of the food additive titanium dioxide (TiO2), but its impact on human health is unknown. The widespread use of food-grade TiO2 (E171) includes commonly consumed products, such as sweets, gums, white salad dressings, dairy creamers, pharmaceutical fillers, and toothpaste. Production of TiO2 in the U.S. is expected to increase more than 8.9% from 2016 to 2025. There are major limitations with current estimations of dietary TiO2 intake in humans. Such limitations include assessing TiO2 content solely from white-colored foods and including only foods with TiO¬2 labeled as such on its packaging. Natural food products, however, may also contribute a substantial amount of TiO¬2 to the diet. There is also a large variation in the estimated ingestion of TiO2 between studies which is likely due to differences in populations and varying food supplies, variability in analytical method used for measuring TiO2, and absence of validated dietary estimation tools to measure oral TiO2 exposure. Therefore, estimation of TiO¬2 dietary intake and gut exposure is needed among a free-living U.S. population of adults with a wide variation of intakes.

Pre-clinical models show that greater TiO2 oral exposure may lead to impaired gut health through changes in gut bacterial content and function. TiO2 has been shown to damage intestinal cells where small doses of TiO2 caused changes in normal activity, but not damage to the cell's genetics. After very small particles of TiO2 are taken up by these intestinal cells, it causes mild toxicity and disruption of the cell's function. In addition, very small particles of TiO2 accumulate in intestinal cells and remodel the cell's community in the small intestine, suggesting these particles may get absorbed into the body's blood and general circulation. These results demonstrate that very small particles of TiO2 causes harmful changes to the intestinal cells, is absorbed by the intestinal cells, and once inside, can cause harmfulness and promote abnormal cellular function. There is an urgent need for studies in humans to determine whether high versus low level exposure to TiO¬2 is related to gut inflammation and disruption in gut function.

The current study will fill these research gaps by testing the hypothesis that long term dietary exposure of TiO2 is related to gut inflammation and disturbs gut bacteria in humans. This hypothesis will be tested for the first time via these specific aims: 1) to quantify dietary TiO2 exposure by estimating dietary intake and measuring the fecal output of TiO2 in 80 adults; 2) to establish the relationship of dietary TiO2 with gut bacteria and their activity; and 3) to determine whether dietary TiO2 exposure is related to gut inflammation and associated inflammatory pathways.

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons between the ages of 18 to 30 y.

Exclusion Criteria:

* <18 years and >30 years
* antibiotic use in the past 6 months
* laxative use in the past 30 days
* self-reported fever, cancer, or gastrointestinal disease (e.g., inflammatory bowel diseases, C. difficile infection
* use of selective serotonin reuptake inhibitors (SSRI's)
* use of non-steroidal anti-inflammatory drugs (NSAIDs) within 10 days
* daily use of proton pump inhibitors
* history of gastrointestinal alteration (e.g., appendectomy, gastric bypass surgery)
* pregnancy.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited from the greater Lowell area, Massachusetts.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-11-28 (Actual)

PRIMARY OUTCOMES:
Gut microbiota taxonomy and expressed pathways | During the study week, three consecutive day period.
  To evaluate the phylogeny and taxonomy of the gut microbiota in each of the three fecal samples per participant, fecal DNA and RNA will be isolated and purified and subject to Illumina-tag PCT to amplify 16S rRNA genes. Samples will be subject to metatranscriptomics sequencing to compare microbial community level expression signatures associated with fecal TiO2.

SECONDARY OUTCOMES:
Concentration of Intestinal Inflammation Biomarkers in Feces | During the study week, three consecutive day period.
  To evaluate intestinal inflammation, the concentrations of fecal calprotectin, lactoferrin, and myeloperoxidase will be measured in stool using Immundiagnostik ELISA kits.
Concentration of Intestinal Homeostasis and Permeability Biomarkers in Feces | During the study week, three consecutive day period.
  To evaluate intestinal homeostasis and permeability, the concentrations of fecal α-1-antitrypsin (AAT) and zonulin will be measured in stool using Immundiagnostik ELISA kits.
Concentration of Intestinal Oxidative Stress Biomarkers in Feces | During the study week, three consecutive day period.
  To evaluate intestinal oxidative stress, the concentrations of leukotriene D4 (LD4) and 3-nitrotyrosine (3-NT) will be measured by liquid chromatography electron spray ionization tandem mass spectrometry (LC-ESIMS/MS).

CONTACTS AND LOCATIONS:
Overall Officials: Kelsey M Mangano, PhD, Principal Investigator — University of Massachusetts, Lowell
Locations (1):
- University of Massachusetts, Lowell, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified data to be released to other researchers upon request to the PI.